CLINICAL TRIAL: NCT04555343
Title: Intravesical Antifibrinolytic for Patients With Hematuria and Clot Retention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: BC Support Unit (Other); Michael Smith Foundation for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHREB 2020-085
Record Dates: First submitted 2020-08-14; First posted 2020-09-18 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Urologic Diseases; Prostate Cancer; Bladder Cancer; Urinary Retention; Hematuria; Nurse Physician Relations; Nurse's Role; Patient Satisfaction
MeSH Terms: conditions — Urologic Diseases; Prostatic Neoplasms; Urinary Bladder Neoplasms; Urinary Retention; Hematuria; Patient Satisfaction | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: convenience sampling of patients presenting to the emergency, all receiving intervention, no blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention- TXA (Experimental): Drug: one-time intravesical administration of 1gm of TXA instilled via urinary catheter, instilled for 15min before continuous bladder irrigation treatment beings.
  1gm of TXA will be mixed with 100cc NS
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — 1gm instilled instravesically
  Other Names: TXA

SUMMARY:
A study looking at the feasibility of doing a full-scale RCT that investigates the use of tranexamic acid intravesically prior to continuous bladder irrigation treatment in the emergency department for urinary retention due to clots.

We want to know:

* patient experience and acceptability of the intervention
* study procedures (recruitment, site appropriateness, staff engagement)
* safety data
* identify resource use

DETAILED DESCRIPTION:
Urinary retention due to high clot burden is a common and resource-intensive condition. Patients who have recently had prostate surgery or who have bladder cancer can often present with urinary retention due to clots. Currently, the standard treatment for hematuria and clot retention that has led to urinary retention is continuous bladder irrigation (CBI) treatment.

CBI treatment is a nursing intensive procedure that is associated with lengthy hospital stays for the patient. CBI treatment is a catheter inserted into the urethral opening that allows a continuous flow of irrigation fluid into and out of the bladder. Initial manual irrigation of clots is also a part of the standard of care. Catheter insertion is a painful procedure, and there is distress during treatment as patients are confined to bed and experience discomfort related to the catheter blockage. CBI treatment may be discontinued as the urine clears of blood only to have it restarted as new clots form. CBI treatment requires a high level of nursing resources as the irrigation fluid must be regularly changed and removed. It also tends to require multiple episodes of manual irrigation by the nurse when it becomes blocked. The procedure is not only distressing and invasive for the patient, but also takes away resources from other patients. The procedure is labor intensive for nursing staff as it requires constant monitoring and frequent episodes of lengthy manual clot irrigation resulting in nursing resource strain and neglect of other patients.

There has been recent interest in adding antifibrinolytics, such as tranexamic acid (TXA), to the standard treatment protocol to stop hematuria and clot retention and thereby decrease patient and staff burden and improve outcomes. TXA is a synthetic lysine analog that prevents the breakdown of clots and facilitates clot stabilization to promote tissue healing. It intervenes at the end of the coagulation pathway to promote clot stabilization. The bladder and prostate are prone to clot breakdown and therefore hematuria, as their tissue naturally promotes clot breakdown. For this reason, TXA has been used extensively in urological surgeries to prevent bleeding complications and has demonstrated effectiveness with an excellent safety profile.

Historically, TXA was given either orally, intramuscularly, or intravenously. However, there is increasing interest in using TXA topically due to a decreased systemic absorption of TXA compared to oral or intravenous use. Our team is interested in exploring the effect TXA has when administered intravesically - i.e., instilled directly into the bladder. Specifically, we are proposing the use of TXA directly into the bladder to obtain preliminary data about the effects on the clinical course of patients requiring CBI treatment for hematuria and clot retention.

Intervention:

A 22-24F three-way Foley catheter will be inserted as per standard nursing protocols, and the treating nurse will manually irrigate the bladder to remove as many clots as possible upon catheter insertion before TXA instillation. One gram of TXA will be mixed with 100 ml of normal saline, then directly instilled into the bladder via the catheter. The catheter will be clamped with the medication in-situ for 15 minutes to allow the medication to have sufficient time in contact with the bladder tissue. After 15 minutes, the catheter will be unclamped, and CBI treatment will be carried out as per standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* complaint of hematuria or urinary retention
* requiring CBI treatment
* able to consent to the study.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Use of anticoagulants (warfarin, heparin, DOACs, etc.)
* known coagulopathy (genetic bleeding disorders, acquired deficiencies)
* urinary tract infection or pyelonephritis
* known hypersensitivity to TXA
* known renal failure
* known or history of thrombosis/thromboembolism (retinal vein/artery occlusion, deep vein thrombosis, pulmonary embolism)
* cognitive impairment rendering unable to provide informed consent and not having a substitute decision-maker present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of study procedures to participants as assessed by successful consenting retention | 20 patients total or a maximum of six months
  measured by the number of eligible patients and number that consent to the study intervention
Participant recruitment time as measured by the time between identification of patient to consent completion | 20 patients total or a maximum of six months
  Patient triage time will be compared to time consent was obtained
Times to intervention- measured by time from consent to time intervention initiated | 20 patients total or a maximum of six months
  all participants will have consent and intervention time documented

SECONDARY OUTCOMES:
Trial site appropriateness as measured by total number of participants recruited within study time | 20 patients total or a maximum of six months
  Both sites will document total number of patients recruited within study time
Incidence of treatment emergent adverse events as assessed by the CTCAE v3.0 severity scale | 20 patients total or a maximum of six months
  All participants will be followed throughout their hospital admission and all adverse events will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Abdalvand, MD, Principal Investigator — Fraser Health Authority
Locations (2):
- Canada (2):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Eagle Ridge Hospital, Port Moody, British Columbia

IPD SHARING:
Plan to Share IPD: No